CLINICAL TRIAL: NCT06755788
Title: Effects of Intraoperative Glycemic Management Strategies Assisted with RT-CGM on TIR and Postoperative Recovery During Pancreaticoduodenectomy: a Randomized Controlled Trial
Brief Title: Effects of Intraoperative Glycemic Management Strategies Assisted with RT-CGM on TIR and Postoperative Recovery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2023-I2M-CT-B-028
Record Dates: First submitted 2024-12-17; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Continuous Glucose Monitoring
Keywords: glycemic management; pancreaticoduodenectomy; time in range

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study is blinded to participants; however, it is not feasible to blind the surgeons and anesthesiologists. The outcome assessors remain blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RT-CGM (Experimental): Intraoperative blood glucose monitoring and management based on a real-time RT-CGM system.
  Interventions: Device: RT-CGM
- Control (Other): Patients enrolled in the control group will have the CGM sensor attached the day before surgery but the CGM , interstitial glucose readings, and alerts will be masked during the operation.
  Interventions: Device: Control

INTERVENTIONS:
Device: RT-CGM — In the RT-CGM group, patients will wear a CGM sensor the day before surgery. Before entering the operating room, capillary blood glucose will be measured and compared with CGM interstitial glucose values for calibration. The target range for intraoperative blood glucose management is 3.9-10.0 mmol/L, with arterial blood gas measurements required at least every 2 hours. Following the administration of insulin or glucose, arterial blood gases should be retested at least every hour. RT-CGM monitoring will also be employed during surgery. A tablet in the operating room will be configured with low and high glucose alerts set at 3.9 mmol/L and 10.0 mmol/L, respectively. When an alarm is triggered, arterial blood gases will be rechecked, and glucose levels will be adjusted based on the arterial blood glucose results. If interstitial glucose values do not reach the intervention threshold, arterial blood gas measurements are recommended every 30 minutes.
  Arms: RT-CGM
Device: Control — In the control group, patients will wear a CGM sensor the day before surgery. Before entering the operating room, capillary blood glucose will be measured and compared with CGM interstitial glucose values for calibration. The target range for intraoperative blood glucose management is 3.9-10.0 mmol/L, with arterial blood gas measurements required at least every 2 hours. Following the administration of insulin or glucose, arterial blood gases should be retested at least every hour. CGM monitoring will also be employed during surgery, but the CGM interstitial glucose readings and alerts will be masked during the operation. The final intraoperative glucose management approach will be determined by the anesthesiologist, considering the patient's condition and surgical circumstances. The anesthesiologist can choose the intravenous insulin adjustment protocol we recommend.
  Arms: Control

SUMMARY:
The purpose of this study is to investigate the effect of intraoperative blood glucose management based on real-time continuous glucose monitoring ( RT-CGM) on time in range (TIR) and postoperative recovery during pancreaticoduodenectomy. The primary outcome is intraoperative TIR. Additionally, it aims to compare the differences in other glucose metrics, quality of postoperative recovery, and 30-day postoperative complications and mortality between the two glycemic management methods .

DETAILED DESCRIPTION:
Pancreaticoduodenectomy (PD) is the standard surgical procedure for treating malignancies of the pancreatic head, distal bile duct, and periampullary region. Due to its extensive scope, high demands for anastomosis, and prolonged operative time, PD is considered one of the most complex surgeries in general surgery. Perioperative management of PD presents unique challenges, particularly in glycemic control. In addition to stress-induced hyperglycemia caused by surgery, Patients with PD are more prone to perioperative glycemic disturbances compared to other surgeries. The main reasons include insulin resistance, resection of pancreatic tissue during surgery, and early postoperative nutritional support. However, perioperative glycemic management guidelines often receive limited attention. Several studies have reported low adherence to recommendations for glycemic monitoring and insulin administration among healthcare professionals. This issue is also evident during the perioperative period of PD, where demanding workloads may lead to neglect of glycemic management, and insulin therapy poses risks of hypoglycemia.

Continuous glucose monitoring (CGM) technology uses subcutaneous electrodes to monitor interstitial glucose levels electronically. RT-CGM provides continuous, comprehensive, and reliable glycemic data, capturing trends and fluctuations in glucose levels, and identifying hidden hyperglycemia and hypoglycemia. It overcomes the limitations of traditional glucose monitoring, such as pain from finger pricks, delayed assessments, and an inability to reflect glucose variability. The latest diabetes guidelines in China and the United States incorporate Time in Range (TIR), derived from CGM, as a new metric for glycemic control. CGM is gradually being used in glycemic management for diabetic patients, and its efficacy and safety have been consistently demonstrated in randomized controlled trials and real-world studies. A randomized controlled trial involving 299 patients with type 2 diabetes showed that CGM improved TIR by 7.9% over 12 months compared to fingerstick glucose monitoring.

Pancreaticoduodenectomy (PD) is the standard surgical procedure for treating malignancies of the pancreatic head, distal bile duct, and periampullary region. Due to its extensive scope, the high demands for anastomosis, and prolonged operative time, PD is considered one of the most complex surgeries in general surgery. Perioperative management of PD presents unique challenges, particularly in glycemic control. In addition to stress-induced hyperglycemia caused by surgery, patients undergoing PD are more susceptible to perioperative glycemic disturbances than those undergoing other types of surgery. The primary factors contributing to this include insulin resistance, the resection of pancreatic tissue during surgery, and early postoperative nutritional support. However, perioperative glycemic management guidelines often receive limited attention, with several studies reporting poor adherence to recommendations for glycemic monitoring and insulin administration among healthcare professionals. This issue is particularly evident during the perioperative period of PD, where heavy workloads may lead to neglect of glycemic management, and insulin therapy may increase the risk of hypoglycemia.

Continuous glucose monitoring (CGM) technology uses subcutaneous electrodes to electronically monitor interstitial glucose levels. Real-time CGM (RT-CGM) provides continuous, comprehensive, and reliable glycemic data, capturing glucose trends and fluctuations while identifying hidden hyperglycemia and hypoglycemia. It overcomes the limitations of traditional glucose monitoring, such as pain from finger pricks, delayed assessments, and an inability to reflect glucose variability. Both China and the United States have incorporated Time in Range (TIR) from CGM data as a key metric for glycemic control in their latest diabetes guidelines. CGM is increasingly used for managing glycemia in diabetic patients, with its efficacy and safety consistently demonstrated in randomized controlled trials and real-world studies. For instance, a randomized controlled trial with 299 patients with type 2 diabetes found that CGM improved TIR by 7.9% over 12 months compared to fingerstick glucose monitoring.

In recent years, the use of CGM has expanded to hospitalized patients, and its adoption is growing in clinical settings. However, compared to medical inpatients and ICU patients, surgical patients rarely use CGM, and studies on its use during surgery are limited. CGM systems measure interstitial glucose every minute and provide real-time alerts for values outside the target range. These alerts help clinicians intervene promptly to manage perioperative hyperglycemia or hypoglycemia, minimizing risks and reducing the burden of traditional blood glucose testing on both patients and medical staff. This study explores the benefits of CGM-assisted glycemic management during PD, promoting dynamic and precise glycemic control during PD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Scheduled for pancreaticoduodenectomy
* ASA classification I-III

Exclusion Criteria:

* Emergency surgery
* scheduled for MRI the day before surgery
* Allergy to CGM sensor
* Communication barriers or refusal to participate
* BMI < 18.5 kg/m²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative time in range (TIR) | during surgery
  Time in range (TIR) from CGM generally refers to the percentage of time that glucose levels stay within a target range (3.9-10 mmol/L)

SECONDARY OUTCOMES:
Intraoperative insulin dosage | during surgery
  unit
Intraoperative time above range (TAR) | during surgery
  Time above range (TAR) from CGM generally refers to the percentage of time glucose levels exceed the upper limit of the target range (>180 mg/dL).
Intraoperative time below range (TBR) | during surgery
  Time below range (TBR) from CGM generally refers to the percentage of time glucose levels fall below the lower limit of the target range (<70 mg/dL).
Intraoperative mean glucose | during surgery
  The average glucose level recorded by the CGM over a specified period
Intraoperative coefficient of variation (CV) | during surgery
  Coefficient of variation (CV) from CGM generally refers to the degree of fluctuation in glucose levels, typically expressed as a percentage of the coefficient of variation.
Postoperative time in range (TIR) | Throughout the 72 hours after surgery
  Time in range (TIR) from CGM generally refers to the percentage of time that glucose levels stay within a target range (3.9-10 mmol/L)
Postraoperative time above range (TAR) | Throughout the 72 hours after surgery
  Time above range (TAR) from CGM generally refers to the percentage of time glucose levels exceed the upper limit of the target range (>180 mg/dL).
Postoperative time below range (TBR) | Throughout the 72 hours after surgery
  Time below range (TBR) from CGM generally refers to the percentage of time glucose levels fall below the lower limit of the target range (<70 mg/dL).
Postoperative mean glucose | Throughout the 72 hours after surgery
  The average glucose level recorded by the CGM over a specified period
Postoperative coefficient of variation (CV) | Throughout the 72 hours after surgery
  Coefficient of variation (CV) from CGM generally refers to the degree of fluctuation in glucose levels, typically expressed as a percentage of the coefficient of variation.
Quality of Recovery-15 score on the third day after surgery | on the third day after surgery
  Using Quality of Recovery-15 questionnaire to evaluate the quality of perioperative recovery. Quality of Recovery-15 consists of 15 comprehensive questions, including physical comfort (5 items), psychological support (2 items), physical independence (2 items), emotional state (4 items), and pain (2 items), each item is scored with 0-10 points, 0 represents poor state, 10 represents good state, and the total score ranging from 0 to 150 is the Quality of Recovery-15 score of the patient. A higher score indicates a better quality of recovery.
The rate of surgery-related complications | 30 days after surgery
  surgery-related complications including clinically relevent postoperative pancreatic fistula,bile leakage,chyle leak,postpancreatectomy hemorrhage,abdominal infection,delayed gastric emptying.
Quality of Recovery-15 score on the 30th day after surgery | on the 30th day after surgery
  Using Quality of Recovery-15 questionnaire to evaluate the quality of perioperative recovery. Quality of Recovery-15 consists of 15 comprehensive questions, including physical comfort (5 items), psychological support (2 items), physical independence (2 items), emotional state (4 items), and pain (2 items), each item is scored with 0-10 points, 0 represents poor state, 10 represents good state, and the total score ranging from 0 to 150 is the Quality of Recovery-15 score of the patient. A higher score indicates a better quality of recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Le Shen, PhD, Principal Investigator — Peking Union Medical College Hospital